CLINICAL TRIAL: NCT03502005
Title: "Efficacy, Safety, and Tolerability of Switching EFV/TDF/FTC to BIC/FTC/TAF in Virologically Suppressed Adults With HIV-1 Infection."
Brief Title: Efficacy, Safety & Tolerability of Switching EFV/TDF/FTC to BIC/FTC/TAF in Virologically Suppressed Adults With HIV-1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Midland Research Group, Inc. (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IN-US-380-4543
Record Dates: First submitted 2018-03-14; First posted 2018-04-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Intervention Model Description: Prospective 48 week single cohort study to evaluate the efficacy and safety of switching from ATRIPLA to BIKTARVY® in HIV-1 infected adult subjects who are virologically suppressed (HIV-1 RNA < 50 copies/mL).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- BIKTARVY® (Experimental): initiation of single pill once daily bictegravir/emtricitabine/tenofovir alafenamide from prior efavirenz/emtricitabine/tenofovir DF
  Interventions: Drug: bictegravir/emtricitabine/tenofovir alafenamide

INTERVENTIONS:
Drug: bictegravir/emtricitabine/tenofovir alafenamide — Discontinue ATRIPLA® and initiate BIKTARVY®
  Other Names: BIKTARVY® (BIC/FTC/TAF)

SUMMARY:
This study evaluates the efficacy, safety and tolerability of switching from the older, established single tablet regimen of ATRIPLA® (EFV/FTC/TDF) to a new single tablet regimen of BIKTARVY® (BIC/FTC/TAF), in HIV-1 infected adult subjects who are virologically suppressed (HIV-1 RNA<50 copies/mL).

DETAILED DESCRIPTION:
Therapeutic dosage of the tenofovir disoproxil fumarate (TDF) component of ATRIPLA® requires plasma concentrations of the drug that are associated with nephrotoxicity and decreased bone mineral density. Tenofovir alafenamide fumarate (TAF) has a unique metabolism that results in higher intracellular levels of the active phosphorylated moiety tenofovir-diphosphate. Compared with TDF, the therapeutic dosage of TAF reduces tenofovir plasma concentrations by over 90%. This reduction in plasma concentration results in decreased renal and bone risks. TAF has the potential to improve on the efficacy and safety profile of TDF.

Efavirenz, another component of ATRIPLA® is widely associated with neuropsychiatric side-effects, including sleep disturbances, depression, and anxiety. Switching from Efavirenz to an integrase inhibitor is associated with improvements in mood.

Bictegravir (BIC) is a novel, once daily integrase inhibitor. It has been shown to have potent antiviral activity, a favorable pharmacokinetic profile, good tolerability and an improved resistance profile when compared to previous integrase inhibitors. In a phase 2 trial investigating previously untreated people with HIV, bictegravir plus emtricitabine and tenofovir alafenamide (BIKTARVY®) vs dolutegravir, plus emtricitabine and tenofovir alafenamide both showed high efficacy up to 24 weeks and both regimens were well tolerated.

Additionally, switching HAART experienced patients to BIKTARVY® has been shown to be non-inferior to continuation of regimens containing Atazanavir or Darunavir, when they were given with either lamivudine/abacavir or FTC/TDF.

The Investigators plan to evaluate in a real world setting the efficacy, safety and tolerability of switching from the older, established single tablet regimen of ATRIPLA® (EFV/FTC/TDF) to a new single tablet regimen of BIKTARVY® (BIC/FTC/TAF).

Within the limitations of a real-world study, Investigators have attempted to replicate the protocol of Gilead Science's Phase 3 study evaluating a switch to BIC/FTC/TAF from dolutegravir plus either FTC/TAF or FTC/TDF14. This will have the potential benefit of comparing different regimen switches as well as potentially adding robustness to the body of data regarding BIC/FTC/TAF.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* On a stable antiretroviral regimen consisting of ATRIPLA® for at least the 6 consecutive months preceding Screening Visit.
* Plasma HIV-1 RNA concentrations at undetectable levels for at least 6 consecutive months prior to the screening visit and have HIV RNA< 50 copies/mL at the Screening Visit.
* Estimated GFR ≥30mL/min according to the Cockcroft-Gault formula for creatinine clearance.
* Hepatic transaminases (AST and ALT) ≤5x upper limit of normal (ULN)
* Total bilirubin ≤1.5 mg/dL, or normal direct bilirubin.
* Adequate hematologic function (hemoglobin ≥ 8.5g/dL; platelets ≥ 50,000/mm3; absolute neutrophil count ≥1,000/mm3)
* Female subjects of reproductive potential using a reliable and consistent method of birth control for at least three months prior to study dosing. Male subjects should use condoms when engaging in intercourse of reproductive potential.
* The ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures.

Exclusion Criteria:

* A new AIDS-defining condition diagnosed within 30 days prior to screening.
* Individuals with decompensated cirrhosis. (i.e. ascites, encephalopathy, etc.)
* Pregnancy
* A history of malignancy within the past 5 years (prior to screening) or ongoing malignancy other than cutaneous Kaposi's sarcoma (KS), basal cell carcinoma, or resected, noninvasive cutaneous squamous carcinoma. Individuals with cutaneous KS are eligible but must not have received any systemic therapy for KS within 30 days prior to baseline.
* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to baseline.
* Life expectancy < 1 year.
* Subject participation in any clinical trial without prior approval from the Investigator.
* Concomitant use of disallowed agents from Table 2
* Participation in any other investigation study 30 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
assess proportion of patients who develop increase in HIV-1 RNA viral load of ≥ 50 copies/mL | 24 weeks
  by week 24

SECONDARY OUTCOMES:
assess stability of kidney function by serial measuring of serum creatinine mg/dL | 48 weeks
  weeks 24 and 48
Assess effect on restoration of immune markers by serial measurement of CD4+ cells | 48 weeks
  weeks 24 and 48
assess effect on lipid cardiovascular risk factors by serial measurement of triglycerides and HDL/LDL cholesterol | 48 weeks
  weeks 24 and 48
assess proportion of patients who continue to have HIV-1 RNA measured <50 copies/mL | 48 weeks
  weeks 24 and 48
Assess patient reported outcomes by two validated patient questionnaires Philadelphia Sleep Quality Index and HIV Symptom Index | 48 weeks
  by week 48
assess patient weight variations from baseline | 48 weeks
  weeks 24 and 48

CONTACTS AND LOCATIONS:
Overall Officials: Noah Lee, DO, Principal Investigator — Midland Research Group, Inc.
Locations (1):
- Midland Research Group, Inc, Oakland Park, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
CROI 2020

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/05/NCT03502005/Prot_SAP_001.pdf
  • Informed Consent Form (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT03502005/ICF_002.pdf